CLINICAL TRIAL: NCT02260479
Title: The Effect of Preheated Skin Disinfection in Relation to Room-temperature Skin Disinfection on Bacterial Colonization During Pace Device Implantation: a Randomized Controlled Non-inferiority Trial.
Brief Title: Preheated Skin Disinfection vs Room-temperature on Bacterial Colonization During Pace Device Implantation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Camilla Wistrand, Operating room nurse, Örebro University, Sweden
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OpPm2013
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Colonization
Keywords: skin disinfection; bacterial colonization; perioperative; chlorehexidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Preheated chlorhexidine (Active Comparator): Preheated skin disinfection with 36ᵒC Chlorhexidine 5mg/ml in 70% alcohol.
  Interventions: Procedure: Preheated
- Room temperature chorhexidine (No Intervention): Room temperature skin disinfection with 20ᵒC Chlorhexidine 5mg/ml in 70% alcohol.

INTERVENTIONS:
Procedure: Preheated — Skin disinfection solution is preheated in a warming cupboard
  Arms: Preheated chlorhexidine

SUMMARY:
The primary aim was to investigate if preheated skin disinfection with Chlorhexidine in alcohol was non-inferior compared to room-temperature regarding skin colonization as well as bacterial colonization in wound, skin temperature and patients experiences.

DETAILED DESCRIPTION:
Patients were randomly assigned to preheated (36ᵒC, intervention) skin disinfection (Chlorhexidine 5mg/ml in 70% alcohol) or room temperature (20ᵒC, control) skin disinfection (Chlorhexidine 5mg/ml in 70% alcohol). Patient´s enrollment to operation was made by an external controller who had no closer knowledge of present study. All patients were asked to participate in that sequence they arrived to the OR department when study nurse was present. Assignment took place directly after patients consent. Patients were stratified into gender and thereafter randomly allocated to preheated or control group, based on a computer-generated randomization list made by an independent statistician. Patients showered, scrubbing their whole body and hair twice with 4% chlorhexidine soap Descutan® (Fresenius Kabi AB, Uppsala, Sweden) prior to surgery. and patients were prepared after skin disinfection with a microbial sealant. Most patients were elective and arrived the morning of surgery to the hospital. Following standard procedures, intravenously administered antibiotic prophylaxis (cloxacillin 2 g) was administrated at the ward 30 minutes before surgery. In the OR the patients wore a disposable cap and were positioned on the operating table. The OR temperature were 19°C with upward displacement ventilation. Sterile disposable surgical gowns (Samutprakarn, Thailand/Mölnlycke Health Care AB, Göteborg, Sweden) and indicator gloves (Selangor, Malaysia/Mölnlycke Health Care AB Göteborg, Sweden) were worn by the surgeon and OR nurse. Other OR staff (n=2) wore cotton scrubs, short-sleeved tunic shirt with cuffs at the arms, and trousers with cuffs at the ankles. They also wore disposable helmets and facemasks. Both groups were given skin disinfection during 2 minutes with the same amount of solution (Chlorhexidine 5mg/ml in 70% alcohol). The skin disinfection (Chlorhexidine 5mg/ml, in alcohol) was stored in room-temperature and was measured to keep 20ᵒC while the preheated was stored in a warming cupboard who kept 36ᵒC. The participants were disinfected from cheek down over sternum according to routine procedures. Sterile material for draping and clothing were for single use only. Cultures were obtained at four occasions using a nylon flocked swab (Copan ESwab, Italia SpA): before skin disinfection on skin surface; after skin disinfection on skin surface; directly after the incision, at completion of the incision, and finally before start of closing sutures. Swab cultures were rubbed for 15 seconds slightly moist with saline on skin surface (incision site). Swabs taken in the wound were rubbed along the inside of the incision for 15 seconds with a dry swab. Surgery was performed by two cardiologists. Cultures were kept cold until arrival at the Department of Laboratory medicine, Clinical Microbiology. Cultures were taken care of and analyzed according to a specific protocol designed especially for the study.

ELIGIBILITY:
Inclusion Criteria:

* could read and understand Swedish

Exclusion Criteria:

* infection in existing implanted device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2013-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Bacterial cultures | perioperative
  Skin cultures (eSwab) taken before and after skin disinfection

SECONDARY OUTCOMES:
Surgical site infections | Three month after surgery
bacterial colonization in wound | perioperative
  Cultures taken in wound at time for incision and before closing sutures
Skin temperature | perioperative
  Skin temperature was taken before and after skin disinfection
Patients experience of skin disinfection | Perioperative
  Numerical rating scale, 0-10 (0=pleasant-10=unpleasant)

REFERENCES:
- [Derived] Wistrand C, Nilsson U, Sundqvist AS. Patient experience of preheated and room temperature skin disinfection prior to cardiac device implantation: A randomised controlled trial. Eur J Cardiovasc Nurs. 2020 Aug;19(6):529-536. doi: 10.1177/1474515119900062. Epub 2020 Feb 7. PMID 32028795